CLINICAL TRIAL: NCT03448523
Title: Evaluation of Right To Play's Positive Child and Youth Development Program: A Cluster Randomised Controlled Trial of a School Play-based Intervention to Prevent Peer Violence and Depression in Hyderabad, Pakistan
Brief Title: Evaluation of Right To Play's Positive Child and Youth Development Program in Middle Schools in Hyderabad, Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council, South Africa (Other)
Collaborators: Aga Khan University (Other); Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC025-8/2015
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Peer Violence; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: open label, randomised, efficacy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right To Play's Positive Child and Youth Development program (Experimental): Behavioural intervention
  Interventions: Behavioral: Right To Play's Positive Child and Youth Development program
- Control (No Intervention): No intervention; intervention to be offered after end line assessment

INTERVENTIONS:
Behavioral: Right To Play's Positive Child and Youth Development program — 1. Right To Play's Red Ball Child Play manual provided for 60 hours per annum for two years
  2. Training of junior leaders
  3. Related play-based activities such as sports days
  4. Quarterly awareness sessions with community groups and parents
  5. Summer camps for children
  6. training of teachers on Right To Play's foundational resources, positive disciplining, and gender and child protection
  Arms: Right To Play's Positive Child and Youth Development program

SUMMARY:
This is a RCT conducted with 1752 children in 40 public middle schools in Hyderabad Pakistan with the goal of evaluating the effectiveness of the international non-governmental organisation Right To Play's Positive Child and Youth Development program on reducing peer violence perpetration and victimisation and child depression in a two arm trial where this intervention is compared to a no intervention arm.

DETAILED DESCRIPTION:
Peer violence is an important violence exposure for young adolescents and has been linked to later perpetration or experience of violence in intimate relationships. It is an obstacle to learning and may impact school students' mental health. Prevention of peer violence requires an intervention that empowers youth and teaches them empathy and stronger social skills. The non-governmental organisation Right To Play operates in 18 countries and has a flagship programme that is used in all countries that has never been subject to most rigorous evaluation. It is a multi-faceted programme that has at its heart an intervention that is delivered throughout the school year in two 35 minute sessions games following activities from the manual Red Ball Child Play that focus on 4 areas of youth development: physical, cognitive, social, and emotional components. These structural activities are designed to improve critical thinking, confidence and resilience. They are complimented by a range of additional activities including junior leader training for selected promising young leaders, week long summary camps, sports days and activities to engage parents and members of the community. The main intervention is delivered by coaches employed by Right To Play and given a 3 week training initially, with subsequent regular refresher engagement. They are supported by junior leaders in the games after junior leader training. Training to teachers on the intervention is also provided.

A two-arm, cluster randomised controlled trial based in middle schools in Hyderabad, Sindh province, Pakistan is evaluating this intervention. It is being conducted in 40 schools, half are boys schools (20) and half (20) girls'. Twenty of the schools have been randomised to the intervention arm and twenty to the control (delayed intervention) arm. The outcomes will be addressed using quantitative methods with data collected from students in Grade 6 at the start of the trial. These measures will be conducted pre-intervention and 12, and 24 month follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* Schools: single sex, public middle schools in Hyderabad; willing to participate and commit time during the school day, twice a week, to the intervention sessions; having an outside playground or indoor space in which games could be played, and 35 or more students in the grade-6 class

School student participants: enrolled in grade 6 in one of the study schools; informed consent from parent and child; able to read the national language Urdu or provincial language Sindhi

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1752 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-03-09 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Peer violence victimisation in the past 4 weeks | assessment 2 years post-baseline
  Mean score on the sixteen questions on peer violence victimisation
Peer violence perpetration in the past 4 weeks | assessment 2 years post-baseline
  Mean score on the sixteen questions on peer violence perpetration
Depression | Over last 2 weeks
  Score on the 28 items Children's Depression Inventory 2 (CDI 2)

SECONDARY OUTCOMES:
School performance | 2 years post baseline
  Mean score on four items asking about performance in reading, writing, maths and Pakistan studies . Responses per item are 1=fail, 2=average, 3=excellent
Days of school missed in last 4 weeks | 2 years post-baseline
  Mean
preparations for marriage | 2 years post baseline
  Based on two questions "have you been promised for marriage' and (if so) 'has your family started other preparation for your marriage?' An affirmative response to the latter will be compared to a negative response combined with the category of students who have not been promised in marriage.
Corporal punishment in the past 4 weeks | 2 years post baseline
  Mean score across the 6 questions
Physical punishment at home in past 4 weeks | 2 years post baseline
  Based on two items with four response categories. The mean score will be calculated.
Gender attitudes (13 items measuring acceptability of spousal violence, girls schooling, male respect for women in decision-making and appropriateness of women's participation) | 2 years post baseline
  Mean score

IPD SHARING:
Plan to Share IPD: No
The data will me made available open access but it will not be individual participant data. The details are still being worked out